CLINICAL TRIAL: NCT07335107
Title: Intravenous Tirofiban After Bridging Therapy for Acute Stroke With Atherosclerotic Large Artery Occlusion (RESCUE-AS): A Multicenter, Randomized, Open Label, Blinded Endpoint Study
Brief Title: Intravenous Tirofiban After Bridging Therapy for Acute Stroke With Atherosclerotic Large Artery Occlusion
Acronym: RESCUE-AS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Liping Liu, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE-AS
Record Dates: First submitted 2026-01-05; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Tirofiban; Large vessel occlusion; Intracranial atherosclerotic disease; bridging treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to the experimental group or control group at a 1:1 ratio. Experimental group: will receive intravenous infusion of tirofiban within 5 minutes after randomization at a dose of 0.4 μg/kg/min for 30 minutes, followed by maintenance infusion via an intravenous microinfusion pump at 0.1 μg/kg/min for 23.5 hours (if tirofiban has already been administered intraoperatively, a continuous intravenous microinfusion pump at 0.1 μg/kg/min will be started directly postoperatively and continued for 24 hours). Tirofiban will be discontinued at 24 hours. Control group: will receive standard medical therapy after bridging treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban Group (Experimental)
  Interventions: Drug: Intravenous Tirofiban
- Control Group (Active Comparator)
  Interventions: Drug: Standard Medical Therapy

INTERVENTIONS:
Drug: Intravenous Tirofiban — Intravenous infusion of tirofiban within 5 minutes after randomization at a dose of 0.4 μg/kg/min for 30 minutes, followed by maintenance infusion via an intravenous microinfusion pump at 0.1 μg/kg/min for 23.5 hours (if tirofiban has already been administered intraoperatively, a continuous intravenous microinfusion pump at 0.1 μg/kg/min will be started directly postoperatively and continued for 24 hours). Tirofiban will be discontinued at 24 hours.
  Arms: Tirofiban Group
Drug: Standard Medical Therapy — standard medical therapy after randomization. The antiplatelet regimen is not restricted.
  Arms: Control Group

SUMMARY:
The investigators propose to assess the efficacy and safety of intravenous tirofiban after bridging therapy (endovascular therapy [EVT] following intravenous Tenecteplase) for acute ischemic stroke due to intracranial atherosclerotic disease related large vessel occlusion (ICAD related LVO). This study will recruit 564 patients from about 50 hospitals in China. Inclusion criteria for the trial are: (1)age ≥18 years old, (2)Pre-mRS 0-2, (3)Baseline NIHSS 6-30 points, (4) Baseline ASPECTS ≥6 points, (5) Baseline CTA/MRA diagnosed: the ICA or MCA-M1/M2 occlusion, (6) Receiving bridging therapy (EVT following IV Tenecteplase) within 24 hours from stroke onset (7) Baseline DSA diagnosed: ICAD related LVO(if any one the following criteria is fulfilled: 1) absence of atrial fibrillation; 2) truncal-type occlusion; 3) residual stenosis ≥30% on DSA after the first retriever; 4) researchers determined it to be ICAD-related LVO based on the TOAST classification, (8) Have achieved successful reperfusion after EVT (mTICI ≥2b). Patients with previously known permanent, persistent, or paroxysmal atrial fibrillation, permanent stenting during EVT, severe bleeding or had a higher bleeding risk in the last 6 months, imaging examination before randomization showed the Heidelberg hemorrhage type 1c, 2, or 3 ICH with or without clinical exacerbation, infarct area greater than 50% of the middle cerebral artery blood supply area or infarct volume ≥70ml, cerebral hernia signs, and some other severe organic diseases and an expected survival time of less than 90 days, severe liver insufficiency or renal insufficiency will be excluded. Patients will be randomly assigned to the experimental group or control group at a 1:1 ratio. Experimental group will receive intravenous tirofiban of a dose of 0.4 μg/kilo/min for 30 minutes after the completion of bridging therapy, followed by a continuous infusion of 0.1 μg/kilo/min for up to 24 hours. Then the patient will transition to standard medical therapy, with no restrictions on the antiplatelet regimen but is advised to receive loading dose dual antiplatelet therapy (oral aspirin 100 mg and clopidogrel 300 mg four hours before the end of intravenous tirofiban and daily oral aspirin 100 mg and clopidogrel 75 mg for 30 days). Control group will receive standard medical therapy after bridging treatment. The primary endpoint is the proportion of modified Rankin Scale (mRS) score 0 to 2 at 90±7 days after onset. The primary safety outcome is the symptomatic intracerebral hemorrhage (sICH) within 48 hours after randomization according to ECASS III criteria. This trial will provide important information for the standardization of antiplatelet medication regimens after bridging therapy for improving functional outcomes in patients with acute large vessel atherosclerotic occlusive ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Pre-mRS 0-2.
3. Baseline NIHSS 6-30 points.
4. Baseline ASPECTS ≥6 points.
5. Baseline CTA/MRA diagnosed: the ICA or MCA-M1/M2 occlusion.
6. Receiving bridging therapy (EVT following IV Tenecteplase) within 24 hours from stroke onset.
7. Baseline DSA diagnosed: ICAD related LVO.

   * ICAD-related LVO is assumed if any one the following criteria is fulfilled: (1) absence of atrial fibrillation; (2) truncal-type occlusion; (3) residual stenosis ≥30% on DSA after the first retriever; (4) researchers determined it to be ICAD-related LVO based on the TOAST classification.
8. Patients have achieved successful reperfusion after EVT (mTICI ≥2b).
9. Patients or their eligible surrogates provided informed consent.

Exclusion Criteria:

1. Previously known permanent, persistent, or paroxysmal atrial fibrillation.
2. Permanent stenting during EVT;
3. Patient had severe bleeding or the following conditions, such as active gastrointestinal ulcer, aortic dissection, platelet count <100 ×109/L, hemoglobin <100 g/L, INR≥1.7 in the last 6 months.
4. Contraindication to glycoprotein IIb/IIIa inhibitors.
5. Imaging examination (Flat-panel NCCT/DCT) before randomization showed the following: Heidelberg hemorrhage type 1c, 2, or 3 ICH with or without clinical exacerbation (an increase of ≥4 points in the NIHSS score from baseline or an increase of ≥2 points in any of the NIHSS scores or resulting in intubation, decompression of bone valves, ventricular drainage, or other significant medical/surgical intervention), infarct area greater than 50% of the middle cerebral artery blood supply area or infarct volume ≥70ml, cerebral hernia signs.
6. Vascular malformations, arterial dissection, intracranial aneurysms, tumors (except for small meningiomas), cerebrovascular inflammation, cerebral amyloid angiopathy, or other major non-ischemic craniocerebral diseases (e.g. multiple sclerosis) as diagnosed by head imaging.
7. Acute renal failure, dialysis, or estimated glomerular filtration rate (eGFR) < 30ml/min/1.72m2, or serum creatinine > 220mmol/L (2.5mg/dl).
8. History of severe liver disease, or aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) and/or glutamyltransferase (GGT) ≥3×ULN and/or total bilirubin (TBIL) ≥2×ULN.
9. Acute ST elevation myocardial infarction (MI), acute decompensated heart failure, QTc>500 ms, hospitalization or involuntary coronary intervention due to acute coronary syndrome, MI, cardiac arrest within the past 3 months.
10. Severe non-cardiovascular comorbidity with life expectancy < 3 months (e.g., malignant tumors).
11. Any clinical conditions determined by the study team that may limit adherence to the study process.
12. Currently receiving an investigational drug or device.
13. Women of childbearing age not practicing reliable contraception who do not have a documented negative pregnancy test.
14. The subject's informed consent was not obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of mRS score 0 to 2 | at 90±7 days after onset
  The modified Rankin scale is a measure of disability, with scores ranging from 0 (no symptoms) to 6 (death), with 0 indicating no symptoms at all; 1 indicating no significant disability despite symptoms: able to carry out all usual duties and activities, 2 indicating slight disability: unable to carry out all previous activities but able to look after own affairs without assistance.
symptomatic intracerebral hemorrhage according to ECASS III criteria | within 48 hours after randomization

SECONDARY OUTCOMES:
Ordinal mRS score | at 90±7 days after onset
  The modified Rankin scale is a measure of disability, with scores ranging from 0 (no symptoms) to 6 (death), with 0 indicating no symptoms at all; 1 indicating no significant disability despite symptoms: able to carry out all usual duties and activities, 2 indicating slight disability: unable to carry out all previous activities but able to look after own affairs without assistance; 3 indicating moderate disability: requiring some help, but able to walk without assistance; 4 indicating moderately severe disability: unable to walk without assistance, and unable to attend to own bodily needs without assistance; 5 indicating severe disability: bedridden, incontinent, and requiring constant nursing care and attention; and 6 indicating death.
mRS score 0 to 1 | at 90±7 days after onset
  The modified Rankin scale is a measure of disability, with scores ranging from 0 (no symptoms) to 6 (death), with 0 indicating no symptoms at all; 1 indicating no significant disability despite symptoms: able to carry out all usual duties and activities.
mRS score 0 to 3 | at 90±7 days after onset
  The modified Rankin scale is a measure of disability, with scores ranging from 0 (no symptoms) to 6 (death), with 0 indicating no symptoms at all; 1 indicating no significant disability despite symptoms: able to carry out all usual duties and activities, 2 indicating slight disability: unable to carry out all previous activities but able to look after own affairs without assistance; 3 indicating moderate disability: requiring some help, but able to walk without assistance.
Early reocclusion | within 48±12 hours after randomization
Severe bleeding according to GUSTO criteria | within 48±12 hours after randomization
Early neurological deterioration (increase in NIHSS score ≥4 points within 72 hours after randomization) | within 72±12 hours after randomization
Any intracerebral hemorrhage | within 48±12 hours after randomization
Mortality | within 90 days after onset

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. Sharing IPD will require IRB approval from Tiantan Hospital and other participating institutes in China.

REFERENCES:
- [Result] Zhao W, Che R, Shang S, Wu C, Li C, Wu L, Chen J, Duan J, Song H, Zhang H, Ling F, Wang Y, Liebeskind D, Feng W, Ji X. Low-Dose Tirofiban Improves Functional Outcome in Acute Ischemic Stroke Patients Treated With Endovascular Thrombectomy. Stroke. 2017 Dec;48(12):3289-3294. doi: 10.1161/STROKEAHA.117.019193. Epub 2017 Nov 10. PMID 29127270
- [Result] Kellert L, Hametner C, Rohde S, Bendszus M, Hacke W, Ringleb P, Stampfl S. Endovascular stroke therapy: tirofiban is associated with risk of fatal intracerebral hemorrhage and poor outcome. Stroke. 2013 May;44(5):1453-5. doi: 10.1161/STROKEAHA.111.000502. Epub 2013 Mar 5. PMID 23463755
- [Result] Zi W, Song J, Kong W, Huang J, Guo C, He W, Yu Y, Zhang B, Geng W, Tan X, Tian Y, Liu Z, Cao M, Cheng D, Li B, Huang W, Liu J, Wang P, Yu Z, Liang H, Yang S, Tang M, Liu W, Huang X, Liu S, Tang Y, Wu Y, Yao L, Shi Z, He P, Zhao H, Chen Z, Luo J, Wan Y, Shi Q, Wang M, Yang D, Chen X, Huang F, Mu J, Li H, Li Z, Zheng J, Xie S, Cai T, Peng Y, Xie W, Qiu Z, Liu C, Yue C, Li L, Tian Y, Yang D, Miao J, Yang J, Hu J, Nogueira RG, Wang D, Saver JL, Li F, Yang Q; RESCUE BT2 Investigators. Tirofiban for Stroke without Large or Medium-Sized Vessel Occlusion. N Engl J Med. 2023 Jun 1;388(22):2025-2036. doi: 10.1056/NEJMoa2214299. PMID 37256974
- [Result] RESCUE BT Trial Investigators; Qiu Z, Li F, Sang H, Luo W, Liu S, Liu W, Guo Z, Li H, Sun D, Huang W, Zhang M, Zhang M, Dai W, Zhou P, Deng W, Zhou Z, Huang X, Lei B, Li J, Yuan Z, Song B, Miao J, Liu S, Jin Z, Zeng G, Zeng H, Yuan J, Wen C, Yu Y, Yuan G, Wu J, Long C, Luo J, Tian Z, Zheng C, Hu Z, Wang S, Wang T, Qi L, Li R, Wan Y, Ke Y, Wu Y, Zhu X, Kong W, Huang J, Peng D, Chang M, Ge H, Shi Z, Yan Z, Du J, Jin Y, Ju D, Huang C, Hong Y, Liu T, Zhao W, Wang J, Zheng B, Wang L, Liu S, Luo X, Luo S, Xu X, Hu J, Pu J, Chen S, Sun Y, Jiang S, Wei L, Fu X, Bai Y, Yang S, Hu W, Zhang G, Pan C, Zhang S, Wang Y, Cao W, Yang S, Zhang J, Guo F, Wen H, Zhang J, Song J, Yue C, Li L, Wu D, Tian Y, Yang J, Lu M, Saver JL, Nogueira RG, Zi W, Yang Q. Effect of Intravenous Tirofiban vs Placebo Before Endovascular Thrombectomy on Functional Outcomes in Large Vessel Occlusion Stroke: The RESCUE BT Randomized Clinical Trial. JAMA. 2022 Aug 9;328(6):543-553. doi: 10.1001/jama.2022.12584. PMID 35943471
- [Result] Baek BH, Yoon W, Lee YY, Kim SK, Kim JT, Park MS. Intravenous Tirofiban Infusion After Angioplasty and Stenting in Intracranial Atherosclerotic Stenosis-Related Stroke. Stroke. 2021 May;52(5):1601-1608. doi: 10.1161/STROKEAHA.120.033551. Epub 2021 Apr 1. PMID 33793319
- [Result] Wu C, Sun C, Wang L, Lian Y, Xie N, Huang S, Zhao W, Ren M, Wu D, Ding J, Song H, Wang Y, Ma Q, Ji X. Low-Dose Tirofiban Treatment Improves Neurological Deterioration Outcome After Intravenous Thrombolysis. Stroke. 2019 Dec;50(12):3481-3487. doi: 10.1161/STROKEAHA.119.026240. Epub 2019 Oct 1. PMID 31570084
- [Result] Gao F, Tong X, Jia B, Wei M, Pan Y, Yang M, Sun D, Nguyen TN, Ren Z, Demiraj F, Yao X, Xu C, Yuan G, Wan Y, Tang J, Wang J, Jiang Y, Wang C, Luo X, Yang H, Shen R, Wu Z, Yuan Z, Wan D, Hu W, Liu Y, Jing P, Wei L, Zheng T, Wu Y, Yang X, Sun Y, Wen C, Chang M, Yin B, Li D, Duan J, Sun D, Guo Z, Xu G, Wang G, Wang L, Wang Y, Jia W, Ma G, Huo X, Mo D, Ma N, Liu L, Zhao X, Wang Y, Fiehler J, Wang Y, Miao Z. Bailout intracranial angioplasty or stenting following thrombectomy for acute large vessel occlusion in China (ANGEL-REBOOT): a multicentre, open-label, blinded-endpoint, randomised controlled trial. Lancet Neurol. 2024 Aug;23(8):797-806. doi: 10.1016/S1474-4422(24)00186-8. Epub 2024 Jun 21. PMID 38914085
- [Result] Yang X, Sun D, Huo X, Raynald R, Jia B, Tong X, Wang A, Ma N, Gao F, Mo D, Miao Z; ANGEL-ACT study group. Futile reperfusion of endovascular treatment for acute anterior circulation large vessel occlusion in the ANGEL-ACT registry. J Neurointerv Surg. 2023 Dec 21;15(e3):e363-e368. doi: 10.1136/jnis-2022-019874. PMID 36693725
- [Result] Zhou T, Yi T, Li T, Zhu L, Li Y, Li Z, Wang M, Li Q, He Y, Yang P, Zhang Y, Li Z, Zhang Y, Ye X, Chen W, Wang S, Liu J; DIRECT-MT Registry Investigators. Predictors of futile recanalization in patients undergoing endovascular treatment in the DIRECT-MT trial. J Neurointerv Surg. 2022 Aug;14(8):752-755. doi: 10.1136/neurintsurg-2021-017765. Epub 2021 Sep 2. PMID 34475255
- [Result] Ma Q, Li R, Wang L, Yin P, Wang Y, Yan C, Ren Y, Qian Z, Vaughn MG, McMillin SE, Hay SI, Naghavi M, Cai M, Wang C, Zhang Z, Zhou M, Lin H, Yang Y. Temporal trend and attributable risk factors of stroke burden in China, 1990-2019: an analysis for the Global Burden of Disease Study 2019. Lancet Public Health. 2021 Dec;6(12):e897-e906. doi: 10.1016/S2468-2667(21)00228-0. PMID 34838196
- [Result] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Result] Fu Z, Xu C, Liu X, Wang Z, Gao L. Safety and Efficacy of Tirofiban in Acute Ischemic Stroke Patients Receiving Endovascular Treatment: A Meta-Analysis. Cerebrovasc Dis. 2020;49(4):442-450. doi: 10.1159/000509054. Epub 2020 Jul 30. PMID 32731250
- [Result] Sang H, Xie D, Tian Y, Nguyen TN, Saver JL, Nogueira RG, Wu J, Long C, Tian Z, Hu Z, Wang T, Li R, Ke Y, Zhu X, Peng D, Chang M, Li L, Ruan J, Wu D, Zi W, Yang Q, Li F, Qiu Z. Association of Tirofiban With Functional Outcomes After Thrombectomy in Acute Ischemic Stroke Due to Intracranial Atherosclerotic Disease. Neurology. 2023 May 9;100(19):e1996-e2006. doi: 10.1212/WNL.0000000000207194. Epub 2023 Mar 20. PMID 36941074
- [Result] Yang M, Huo X, Miao Z, Wang Y. Platelet Glycoprotein IIb/IIIa Receptor Inhibitor Tirofiban in Acute Ischemic Stroke. Drugs. 2019 Apr;79(5):515-529. doi: 10.1007/s40265-019-01078-0. PMID 30838514
- [Result] Jovin TG, Nogueira RG, Lansberg MG, Demchuk AM, Martins SO, Mocco J, Ribo M, Jadhav AP, Ortega-Gutierrez S, Hill MD, Lima FO, Haussen DC, Brown S, Goyal M, Siddiqui AH, Heit JJ, Menon BK, Kemp S, Budzik R, Urra X, Marks MP, Costalat V, Liebeskind DS, Albers GW. Thrombectomy for anterior circulation stroke beyond 6 h from time last known well (AURORA): a systematic review and individual patient data meta-analysis. Lancet. 2022 Jan 15;399(10321):249-258. doi: 10.1016/S0140-6736(21)01341-6. Epub 2021 Nov 11. PMID 34774198
- [Result] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Result] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Result] de Havenon A, Zaidat OO, Amin-Hanjani S, Nguyen TN, Bangad A, Abbasi M, Anadani M, Almallouhi E, Chatterjee R, Mazighi M, Mistry EA, Yaghi S, Derdeyn CP, Hong KS, Kvernland A, Leslie-Mazwi TM, Al Kasab S. Large Vessel Occlusion Stroke due to Intracranial Atherosclerotic Disease: Identification, Medical and Interventional Treatment, and Outcomes. Stroke. 2023 Jun;54(6):1695-1705. doi: 10.1161/STROKEAHA.122.040008. Epub 2023 Mar 20. PMID 36938708